CLINICAL TRIAL: NCT02883374
Title: Chidamide for Advanced Cephalic and Cervical Adenocystic Carcinoma: Evaluation of Efficiency and Safety
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dong mei (Other)
Responsible Party: Sponsor-Investigator, Dong mei, Doctor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CancerIHCAMS16-053/1132
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Adenocystic Carcinoma
Keywords: cephalic and cervical adenocystic Carcinoma; Chidamide
MeSH Terms: conditions — Carcinoma, Adenoid Cystic | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chidamide (Experimental): Patients of advanced cephalic and cervical adenocystic carcinoma are given Chidamide 30mg,biw, then the efficacy and safety will be accessed.
  Interventions: Drug: Chidamide

INTERVENTIONS:
Drug: Chidamide
  Other Names: epidaza

SUMMARY:
The purpose of this trial is to evaluate the efficiency and safety of Chidamide in advanced cephalic and cervical adenoid cystic carcinoma. Chidamide is given to patients with advanced cephalic and cervical adenoid cystic carcinoma with the dosage of 30mg,twice a week, then overall survival, event-free survival are accessed for efficiency, and laboratory tests about the function of vital organs are accessed for safety.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of advanced cephalic and cervical adenocystic carcinoma with pathological and imaging evidences, with local relapse or metastasis or refractory towards treatment.
2. Age 18-75, male or female, expected survival≥ 3 months.
3. ECOG 0-2.
4. With at least one evaluable disease focus.
5. Organ functions should fit the following:

Liver: Total bilirubin ≤ 1.5 times of the normal maximum, ALT and AST≤ 2.5 times of the normal maximum. (ALT/AST≤ 5 times of the normal maximum for patients with infiltrative liver disease) Kidney: Serum creatinine ˂ 1.5 folds of the normal maximum; creatinine clearance rate ≥50ml/min (calculated by Cockroft-Gault10 formula)

Exclusion Criteria:

1. History of HDACI treatment.
2. Women during pregnancy or lactation.
3. Patients with a second primary tumor ( this does not include non-melanoma skin cancer received systemic treatment, cured cervical carcinoma in situ of the uterus, or other tumors that have been cured with disease free survival˃ 5 years)
4. Patients with central nervous system defects or mental disorders.
5. Other diseases or contraindications: History of heart disease within 6 months prior to inclusion, including NYHA III-IV heart failure after treatment, coronary heart disease, angina pectoris, myocardial infarction, degree II or III atrioventricular block, severe arrhythmias that need medical treatment, uncontrolled hypertension; liver cirrhosis (Child-Pugh B or C); active infection that has not been controlled, and other conditions that may make the patient unable to complete the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-11; Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Disease control rate | through study completion, an average of 33 months
  percentage of patients who get complete remission, partial remission and stable disease.

SECONDARY OUTCOMES:
Toxicities | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 33 months
  Hematologic toxicities and non-hematologic toxicities including nausea，vomiting，liver, heart and other organ disfunctions.
QOL score | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 33 months
  improvement of patients' feeling and quality of daily life

CONTACTS AND LOCATIONS:
Overall Officials: Mei Dong, Doctor, Principal Investigator — Cancer Hospital Chinese Academy of Medical Science
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Science, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
The data of the trial would be accessable on the corresponding website after the trial has been finished.